CLINICAL TRIAL: NCT03633994
Title: Heparin Intraoperative Instillation for Lower Urinary Tract Symptoms After Benign Hysterectomy: A Randomized Controlled Trial
Brief Title: Heparin Intraoperative Instillation for Lower Urinary Tract Symptoms After Benign Hysterectomy
Acronym: HILUTS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Christ Hospital (Other)
Responsible Party: Principal Investigator, Hyde Yuen, Female Pelvic Medicine and Reconstructive Surgery Fellow, The Christ Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TCH #18-12
Record Dates: First submitted 2018-08-13; First posted 2018-08-16 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Lower Urinary Tract Symptoms; Postoperative Urinary Tract Infection
Keywords: Randomized controlled trial; Heparin instillation
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Heparin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heparin Bladder Instillation (Experimental): At the completion of the scheduled benign hysterectomy, intravesicular bladder instillation containing 40,000U of heparin (40mL of 10,000U heparin/10mL) will be administered be introduced in a retrograde fashion by gravity via Foley catheter. The Foley catheter will be clamped for 30 minutes approximately 1cm from the vaginal opening.
  Interventions: Drug: Heparin
- Normal Saline Bladder Instillation (Placebo Comparator): Patients randomized to the control group will undergo intravesical instillation with 40mL of normal saline. The Foley catheter will be clamped for 30 minutes approximately 1cm from the vaginal opening.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Heparin — Heparin is a readily available glycosaminoglycan (GAG) chemically similar to hyaluronic acid and chondroitin sulfate that is currently used to treat chronic painful bladder or interstitial cystitis. Heparin intravesical treatment is an inexpensive second-line treatment for chronic painful bladder, characterized by urinary frequency, urgency and pain. Heparin has been shown to re-establish the bladder urothelial GAG layer and as already noted was shown to reduce recurrent urinary tract infections by 50%.
  Arms: Heparin Bladder Instillation
Drug: Normal saline — Normal saline bladder instillation
  Arms: Normal Saline Bladder Instillation

SUMMARY:
This study will explore the application of placing heparin into the bladder via a catheter to decrease postoperative lower urinary tract symptoms (LUTS) and urinary tract infection (UTI) symptoms such as urinary frequency, urinary urgency, pain with urination, or difficulty voiding following hysterectomy (surgically removing the uterus). The investigators hypothesize that heparin bladder instillations will reduce LUTS, UTI symptoms, and improve patient satisfaction following hysterectomy.

DETAILED DESCRIPTION:
Data Collection

Subject demographics and history information will be obtained from The Christ Hospital Medical Center's electronic medical record. In addition, preoperative diagnosis, postoperative diagnosis, procedure performed, total operative time, estimated blood loss, intraoperative complications, anterior prolapse repair, use of cystoscopy, preoperative urinalysis, postoperative complications, uterine size, and any urine cultures collected within the 2 week postoperative period will also obtained from the electronic medical record.

The post-operative lower urinary tract symptoms assessments will be collected, the paper records will be secured in a locker labeled with the study identification number, which will then be entered into EXCEL on a password secured database and the paper copy will be disposed of in the secure destruction station.

Descriptive Analysis

Simple statistics and demographics will be done across the two cohorts. Categorical variables will be analyzed using Chi-square while continuous variables (e.g. UTISA scores) will be analyzed using t-test so long as the distribution of the data are normal. Additional analyzes as appropriate will be done to identify group differences based on patient demographics (e.g. age, concomitant procedures, surgeon, estrogen use, foley catheter placement, etc).

Data Analysis and Data Monitoring

The UTISA survey and VAS pain scale both result a continuous variable that between the two cohorts will be compared using a t-Test provided the results distribution is normal. Antibiotic use or self-reported UTI rates are nominal variables that across the cohorts would be compared using a X2.

Data analysis will be performed using statistical software (JMP 13.2.0, SAS Institute Inc., Cary NC, USA). The data will be assembled into a password protected EXCEL (Microsoft, Redmond WA, USA) spreadsheet. A separate password protected spreadsheet will link the study ID and the enrolled patient's MRN. Analysis would be done only on the de-identified data.

Data Storage and Confidentiality

Study data will be managed in a password-protected EXCEL (Microsoft, Redmond WA, USA) spreadsheet on a password-protected computer. A separate password protected spreadsheet linking the study ID and MRN will be kept on a separate password-protected secure drive. This "key" file will be securely destroyed when the data has been fully analyzed. Paper records including consent will be in a locked research drawer, in the designated locked office. The investigators will dispose of any paper documents after data has been analyzed using the CINTAS Secure Destruction Station.

Sample Size

The symptom with the highest sensitivity and specificity to predict a UTI is dysuria. A study in 2013 demonstrated a 50% reduction in UTIs among heparin treated patients, the investigators estimated an effect size of 0.6, assuming mean UTISA dysuria scores of 2 and 1 among the untreated and treated cohorts assessed on post-operative day 1. Assuming an α of 0.05 and 80% power, the investigators estimate requiring 45 subjects per study arm totaling 90 patients. Assuming at least 15% attrition in each arm, the investigators estimate needing to enroll at least 52 patients per study arm to a total of 104 patients.

Plans for recruitment of subjects

No advertisement will be used. The recruitment will take at the time of surgical consent, via phone after patient is identified at the time of preoperative visit, or on the day of surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85-years old
* scheduled to undergo a benign hysterectomy

Exclusion Criteria:

* non-English speakers
* current use of anticoagulants or thrombolytic agents
* known adverse reaction or hypersensitivity to heparin
* history of or active genitourinary tract cancer (bladder, uterine, cervical, ovarian or vaginal)
* history of neurogenic bladder
* pelvic irradiation
* chemical cystitis
* pregnancy
* antibiotic use within the past 30 days
* Surgical procedures involving: anterior or posterior colporrhaphy, vaginal mesh excision, fistula repair, diverticulum repair, urethral reconstruction, planned or incidental cystotomy

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients undergoing benign hysterectomy
Enrollment: 104 (Estimated)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Lower urinary tract symptoms | Postoperative day 14
  lower urinary tract symptoms such as urgency, frequency, dysuria, and hematuria measured by the Urinary Tract Infection Symptoms Assessment Questionnaire (UTISA)

SECONDARY OUTCOMES:
Postoperative antibiotic use | Postoperative day 1 to 14
  Obtained via phone interview
Postoperative patient satisfaction | Postoperative day 14
  Surgical Satisfaction Questionnaire (SSQ-8) assessment conducted via phone interview

CONTACTS AND LOCATIONS:
Locations (1):
- The Christ Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ablove T, Patankar M, Seo S. Prevention of recurrent urinary tract infections by intravesical administration of heparin: a pilot study. Ther Adv Urol. 2013 Dec;5(6):303-9. doi: 10.1177/1756287213504804. PMID 24294288
- [Result] Albo ME, Richter HE, Brubaker L, Norton P, Kraus SR, Zimmern PE, Chai TC, Zyczynski H, Diokno AC, Tennstedt S, Nager C, Lloyd LK, FitzGerald M, Lemack GE, Johnson HW, Leng W, Mallett V, Stoddard AM, Menefee S, Varner RE, Kenton K, Moalli P, Sirls L, Dandreo KJ, Kusek JW, Nyberg LM, Steers W; Urinary Incontinence Treatment Network. Burch colposuspension versus fascial sling to reduce urinary stress incontinence. N Engl J Med. 2007 May 24;356(21):2143-55. doi: 10.1056/NEJMoa070416. Epub 2007 May 21. PMID 17517855
- [Result] Anand M, Wang C, French J, Isaacson-Schmid M, Wall LL, Mysorekar IU. Estrogen affects the glycosaminoglycan layer of the murine bladder. Female Pelvic Med Reconstr Surg. 2012 May-Jun;18(3):148-52. doi: 10.1097/SPV.0b013e31824b76bd. PMID 22543765
- [Result] Ciani O, Arendsen E, Romancik M, Lunik R, Costantini E, Di Biase M, Morgia G, Fragala E, Roman T, Bernat M, Guazzoni G, Tarricone R, Lazzeri M. Intravesical administration of combined hyaluronic acid (HA) and chondroitin sulfate (CS) for the treatment of female recurrent urinary tract infections: a European multicentre nested case-control study. BMJ Open. 2016 Mar 31;6(3):e009669. doi: 10.1136/bmjopen-2015-009669. PMID 27033958
- [Result] Clayson D, Wild D, Doll H, Keating K, Gondek K. Validation of a patient-administered questionnaire to measure the severity and bothersomeness of lower urinary tract symptoms in uncomplicated urinary tract infection (UTI): the UTI Symptom Assessment questionnaire. BJU Int. 2005 Aug;96(3):350-9. doi: 10.1111/j.1464-410X.2005.05630.x. PMID 16042729
- [Result] Cohen SL, Ajao MO, Clark NV, Vitonis AF, Einarsson JI. Outpatient Hysterectomy Volume in the United States. Obstet Gynecol. 2017 Jul;130(1):130-137. doi: 10.1097/AOG.0000000000002103. PMID 28594764
- [Result] Damiano R, Quarto G, Bava I, Ucciero G, De Domenico R, Palumbo MI, Autorino R. Prevention of recurrent urinary tract infections by intravesical administration of hyaluronic acid and chondroitin sulphate: a placebo-controlled randomised trial. Eur Urol. 2011 Apr;59(4):645-51. doi: 10.1016/j.eururo.2010.12.039. Epub 2011 Jan 18. PMID 21272992
- [Result] Desai VB, Xu X. An update on inpatient hysterectomy routes in the United States. Am J Obstet Gynecol. 2015 Nov;213(5):742-3. doi: 10.1016/j.ajog.2015.07.038. Epub 2015 Jul 28. No abstract available. PMID 26226555
- [Result] Dieter AA, Amundsen CL, Edenfield AL, Kawasaki A, Levin PJ, Visco AG, Siddiqui NY. Oral antibiotics to prevent postoperative urinary tract infection: a randomized controlled trial. Obstet Gynecol. 2014 Jan;123(1):96-103. doi: 10.1097/AOG.0000000000000024. PMID 24463669
- [Result] Elkadry EA, Kenton KS, FitzGerald MP, Shott S, Brubaker L. Patient-selected goals: a new perspective on surgical outcome. Am J Obstet Gynecol. 2003 Dec;189(6):1551-7; discussion 1557-8. doi: 10.1016/s0002-9378(03)00932-3. PMID 14710061
- [Result] Foxman B. Epidemiology of urinary tract infections: incidence, morbidity, and economic costs. Dis Mon. 2003 Feb;49(2):53-70. doi: 10.1067/mda.2003.7. PMID 12601337
- [Result] Gagyor I, Bleidorn J, Kochen MM, Schmiemann G, Wegscheider K, Hummers-Pradier E. Ibuprofen versus fosfomycin for uncomplicated urinary tract infection in women: randomised controlled trial. BMJ. 2015 Dec 23;351:h6544. doi: 10.1136/bmj.h6544. PMID 26698878
- [Result] Generali JA, Cada DJ. Intravesical heparin: interstitial cystitis (painful bladder syndrome). Hosp Pharm. 2013 Nov;48(10):822-4. doi: 10.1310/hpj4810-822. PMID 24421434
- [Result] Giesen LG, Cousins G, Dimitrov BD, van de Laar FA, Fahey T. Predicting acute uncomplicated urinary tract infection in women: a systematic review of the diagnostic accuracy of symptoms and signs. BMC Fam Pract. 2010 Oct 24;11:78. doi: 10.1186/1471-2296-11-78. PMID 20969801
- [Result] Givens CD, Wenzel RP. Catheter-associated urinary tract infections in surgical patients: a controlled study on the excess morbidity and costs. J Urol. 1980 Nov;124(5):646-8. doi: 10.1016/s0022-5347(17)55596-2. PMID 7452793
- [Result] Jackson D, Higgins E, Bracken J, Yandell PM, Shull B, Foster RT Sr. Antibiotic prophylaxis for urinary tract infection after midurethral sling: a randomized controlled trial. Female Pelvic Med Reconstr Surg. 2013 May-Jun;19(3):137-41. doi: 10.1097/SPV.0b013e318285ba53. PMID 23611930
- [Result] Karp NE, Kobernik EK, Kamdar NS, Fore AM, Morgan DM. Length of Catheter Use After Hysterectomy as a Risk Factor for Urinary Tract Infection. Female Pelvic Med Reconstr Surg. 2018 Nov/Dec;24(6):430-434. doi: 10.1097/SPV.0000000000000486. PMID 28914703
- [Result] Lake AG, McPencow AM, Dick-Biascoechea MA, Martin DK, Erekson EA. Surgical site infection after hysterectomy. Am J Obstet Gynecol. 2013 Nov;209(5):490.e1-9. doi: 10.1016/j.ajog.2013.06.018. Epub 2013 Jun 13. PMID 23770467
- [Result] Lakeman MM, van der Vaart CH, Roovers JP; HysVA study group. Hysterectomy and lower urinary tract symptoms: a nonrandomized comparison of vaginal and abdominal hysterectomy. Gynecol Obstet Invest. 2010;70(2):100-6. doi: 10.1159/000297507. Epub 2010 Mar 19. PMID 20299800
- [Result] Ley K, Laudanna C, Cybulsky MI, Nourshargh S. Getting to the site of inflammation: the leukocyte adhesion cascade updated. Nat Rev Immunol. 2007 Sep;7(9):678-89. doi: 10.1038/nri2156. PMID 17717539
- [Result] Lusardi G, Lipp A, Shaw C. Antibiotic prophylaxis for short-term catheter bladder drainage in adults. Cochrane Database Syst Rev. 2013 Jul 3;2013(7):CD005428. doi: 10.1002/14651858.CD005428.pub2. PMID 23824735
- [Result] Nomiya A, Naruse T, Niimi A, Nishimatsu H, Kume H, Igawa Y, Homma Y. On- and post-treatment symptom relief by repeated instillations of heparin and alkalized lidocaine in interstitial cystitis. Int J Urol. 2013 Nov;20(11):1118-22. doi: 10.1111/iju.12120. Epub 2013 Feb 22. PMID 23432185
- [Result] Palsson M, Stjerndahl JH, Granasen G, Lofgren M, Sundfeldt K. Patient-reported lower urinary tract symptoms after hysterectomy or hysteroscopy: a study from the Swedish Quality Register for Gynecological Surgery. Int Urogynecol J. 2017 Sep;28(9):1341-1349. doi: 10.1007/s00192-017-3268-9. Epub 2017 Jan 23. PMID 28116468
- [Result] Parsons CL, Zupkas P, Proctor J, Koziol J, Franklin A, Giesing D, Davis E, Lakin CM, Kahn BS, Garner WJ. Alkalinized lidocaine and heparin provide immediate relief of pain and urgency in patients with interstitial cystitis. J Sex Med. 2012 Jan;9(1):207-12. doi: 10.1111/j.1743-6109.2011.02542.x. Epub 2011 Nov 14. PMID 22082303
- [Result] Pham T, Kenton K, Mueller E, Brubaker L. New pelvic symptoms are common after reconstructive pelvic surgery. Am J Obstet Gynecol. 2009 Jan;200(1):88.e1-5. doi: 10.1016/j.ajog.2008.08.010. Epub 2008 Oct 9. PMID 18845285
- [Result] Qin C, de Oliveira G, Hackett N, Kim JY. Surgical duration and risk of Urinary Tract Infection: An analysis of 1,452,369 patients using the National Surgical Quality Improvement Program (NSQIP). Int J Surg. 2015 Aug;20:107-12. doi: 10.1016/j.ijsu.2015.05.051. Epub 2015 Jun 6. PMID 26054658
- [Result] Shepherd AK, Pottinger PS. Management of urinary tract infections in the era of increasing antimicrobial resistance. Med Clin North Am. 2013 Jul;97(4):737-57, xii. doi: 10.1016/j.mcna.2013.03.006. Epub 2013 Apr 29. PMID 23809723
- [Result] Thakar R, Ayers S, Clarkson P, Stanton S, Manyonda I. Outcomes after total versus subtotal abdominal hysterectomy. N Engl J Med. 2002 Oct 24;347(17):1318-25. doi: 10.1056/NEJMoa013336. PMID 12397189
- [Result] Wald HL, Ma A, Bratzler DW, Kramer AM. Indwelling urinary catheter use in the postoperative period: analysis of the national surgical infection prevention project data. Arch Surg. 2008 Jun;143(6):551-7. doi: 10.1001/archsurg.143.6.551. PMID 18559747